CLINICAL TRIAL: NCT02177721
Title: A Field Study to Evaluate the Clinical Benefit and Safety of Raxibacumab in Patients With Symptomatic Inhalational Anthrax in a Mass Exposure Scenario
Brief Title: Clinical Benefit and Safety of Raxibacumab in Patients With Symptomatic Inhalational Anthrax in a Mass Exposure Scenario
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EBS-RAX-200137a
Record Dates: First submitted 2014-05-15; First posted 2014-06-30 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Infections, Bacterial
Keywords: Raxibacumab; anthrax; anti-toxin
MeSH Terms: conditions — Bacterial Infections; Anthrax | interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Raxibacumab arm (Experimental): This is an open-label, single arm study. The study will be implemented for subjects with symptomatic inhalational anthrax who receive FDA-approved raxibacumab as part of medical treatment of anthrax following a mass exposure scenario.
  Intervention: Sampling of subjects or use of subjects salvaged standard of care samples may be considered for the following assessments (if available/applicable): analysis of antibodies to PA (anti-PA), protective antigen (PA), and lethal factor (LF).
  Interventions: Biological: Sample Collection

INTERVENTIONS:
Biological: Sample Collection — Whenever possible serum samples will be collected from all subjects to determine serum raxibacumab concentrations pre-infusion, and at specific timepoints post-infusion. In the event cerebrospinal fluid (CSF), pleural, ascites, or bronchoalveolar lavage (BAL) fluid are collected for ad hoc clinical laboratory testing, any remaining excess sample will be provided to Sponsor for determination of raxibacumab concentrations.
  Any available serum remaining from ad hoc clinical laboratory specimen collections prior to raxibacumab administration will be provided to Sponsor for measurement of serum PA concentrations. In addition, remaining post raxibacumab dose serum specimens may also be analyzed for lethal factor (LF) levels.

SUMMARY:
This field study is designed such that it may be implemented for any individual with symptomatic inhalational anthrax who has been administered raxibacumab for treatment of anthrax following a mass exposure scenario. This study is designed to describe the clinical effectiveness (including course of illness and survival) and safety profile from patients who are treated with raxibacumab as part of their clinical care following exposure to B. anthracis. Study data and other investigational research will be collected prospectively to the extent possible at pre-specified time points. However, because of the logistical complexities that would likely accompany a mass anthrax event, most data in this study is anticipated to be collected retrospectively. During such a mass anthrax event, scavenged blood samples will be utilized where possible to maximize sample analyses and other investigational parameters. Therefore, both retrospective and prospective data collection are allowed in this protocol in order to maximize the amount of information obtained in subjects who have been administered raxibacumab. This field study will be the first opportunity to collect data on B. anthracis-exposed patients treated with raxibacumab, to better understand the clinical benefit and safety of the drug and to further inform patient care and treatment choices for management of anthrax.

DETAILED DESCRIPTION:
The protocol is a post-marketing requirement from the FDA to evaluate the clinical benefit and safety of raxibacumab administered to patients with symptomatic inhalational anthrax as part of their medical care following a mass exposure scenario to Bacillus anthracis.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic inhalational anthrax linked to an identified mass exposure to B. anthracis.
* Women, including pregnant and lactating women, men, and children of all ages who receive a dose of raxibacumab from the Strategic National Stockpile (SNS) as part of their clinical care for symptomatic inhalational anthrax will be eligible to enroll in this study.
* Patients willing and able to adhere to the procedures stated in the protocol.
* Patients (or legally acceptable representative of minors and unconscious adults) willing and able to give written informed consent/assent (as applicable) to participate in the study.

Exclusion Criteria:

* There are no exclusion criteria for patients enrolling in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2035-05 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate Clinical Benefit of Raxibacumab for Patients with Symptomatic Inhalational Anthrax | Up to Day 29
  Evaluate the clinical benefit of raxibacumab for the treatment of inhalational anthrax disease in a mass exposure scenario such as intentional B. anthracis release during a bioterrorist attack.

SECONDARY OUTCOMES:
Evaluate Safety of Raxibacumab for Patients with Symptomatic Inhalational Anthrax | Up to Day 29
  Evaluate the safety of raxibacumab for the treatment of inhalational anthrax disease in a mass exposure scenario such as intentional B. anthracis release during a bioterrorist attack.

OTHER OUTCOMES:
Evaluate the Clinical Course of Disease | Up to Day 29
  To evaluate the clinical course of the disease in patients with inhalational anthrax disease.

CONTACTS AND LOCATIONS:
Overall Officials: Bojan Drobic, PhD, Study Director — Emergent BioSolutions

IPD SHARING:
Plan to Share IPD: No